CLINICAL TRIAL: NCT01394172
Title: Non-invasive Ventilation Generated by External Chest Pressure in Children
Brief Title: A Novel Method of Non-invasive Ventilation in Children
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00018804
Record Dates: First submitted 2011-07-06; First posted 2011-07-14 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Apnea
Keywords: Tidal Volume; Pediatric; Difficult airway; Ventilation; Airway management
MeSH Terms: conditions — Apnea; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to quantify the tidal volume generated by the pressure release immediately following the application of pressure to the chest.

DETAILED DESCRIPTION:
Airway management in the pediatric population differs from the adult population because of differences in their respiratory physiology and anatomy. For example the oxygen consumption is about three times higher in children as compared to adults; therefore, if there is a problem ventilating a child there is a higher impact on oxygen delivery and oxygen reserve. Current guidelines recommend that in respiratory emergencies where one "cannot ventilate and cannot intubate" that a cricothyroidectomy (insertion of a needle through the cricothyroid membrane in the neck) be performed. This procedure is very invasive and difficult to perform, especially in a small child. Since timing and simplicity are essential to successful airway management it is hypothesized that the investigators could utilize the physiological principles behind breathing to ventilate these children using the release of applied pressure to their chest. During, inspiration, the vertical and transverse dimensions of the thorax are increased, generating a negative pressure between the intrapleural space and the chest wall, allowing for air to be drawn into the lungs. As children have a very compliant rib cage one of the theoretical ways to improve lung inflation is to apply external pressure on the chest. The intrathoracic pressure increases above atmospheric pressure and air preferentially flows out of the lungs according to the pressure gradient. When the pressure is released and the chest recoils passively, a negative intrathoracic pressure is generated, which allows for air to flow into the lungs according to the pressure gradient created. If a sufficient tidal volume is generated by the release of pressure from the chest this could potentially become a simple, non-invasive, life-saving technique in children with difficult airways. By adapting the principles described above, it is possible that tidal volume and therefore, gas exchange can take place on release of the pressure applied to the chest.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients under the age of 18 years old.
* All patients requiring a general anesthetic with an endotracheal tube (whether the patient will be intubated with an endotracheal tube will be decided by the anesthesiologist responsible for the case)
* ASA (American Society of Anesthesiologists Physical Status Classification) I to III

Exclusion Criteria:

* Failure to obtain parental consent or patient assent when appropriate (in general children over 8 years old)
* ASA (American Society of Anesthesiologists Physical Status Classification) IV
* Patients with any cardiac pathology
* Patients with any respiratory pathology
* Patients with any form of chest deformity (examples being pectus excavatum, pectus carinatum, scoliosis)
* Patients who had previous cardiac/thoracic surgery

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This is a prospective, cohort study with a sample size of approximately 100 pediatric patients. The population will be stratified equally into the following age groups: neonate (0-28 days or 44 post-conceptual weeks), infants (>1-12 months), toddlers (>12months-3 years), children (>3-8 years), pre-teen (>8-13 years) and adolescent (>13 years).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-06; Primary Completion 2014-05 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Tidal volume (mL), as displayed by the Draeger Narkomed 6400 Anesthesia Machine, after release of manual chest compression | After induction of general anesthesia and until completion of surgery (within an average time of 30 mins to 4 hours)
  One tidal volume is displayed on the Draeger machine immediately after the manual release of chest compression. This outcome is recorded 3 times in each patient after fast manual compressions (1-2 seconds each), with the process performed while the patient is both bag-mask ventilated and intubated.

SECONDARY OUTCOMES:
Force of compression (kg), as displayed by the Lafayette Manual Muscle Tester, measured during each manual chest compression | after induction of general anesthesia and during surgery (between 30 mins and 4 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Ban Tsui, M.D., M.Sc., Principal Investigator — Department of Anesthesiology and Pain Medicine, University of Alberta; Viv Ip, M.D., Study Director — Department of Anesthesiology and Pain Medicine University of Alberta; Sara Horne, B.Sc.(Hons), Study Director — Department of Anesthesiology and Pain Medicine University of Alberta
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Williams AJ. ABC of oxygen: assessing and interpreting arterial blood gases and acid-base balance. BMJ. 1998 Oct 31;317(7167):1213-6. doi: 10.1136/bmj.317.7167.1213. No abstract available. PMID 9794863
- [Background] Adler SM, Wohl ME. Flow-volume relationship at low lung volumes in healthy term newborn infants. Pediatrics. 1978 Apr;61(4):636-40. PMID 662489
- [Background] Braga MS, Dominguez TE, Pollock AN, Niles D, Meyer A, Myklebust H, Nysaether J, Nadkarni V. Estimation of optimal CPR chest compression depth in children by using computer tomography. Pediatrics. 2009 Jul;124(1):e69-74. doi: 10.1542/peds.2009-0153. PMID 19564271
- [Derived] Tsui BC, Horne S, Tsui J, Corry GN. Generation of tidal volume via gentle chest pressure in children over one year old. Resuscitation. 2015 Jul;92:148-53. doi: 10.1016/j.resuscitation.2015.02.021. Epub 2015 Mar 4. PMID 25749553